CLINICAL TRIAL: NCT00847548
Title: Treatment of Intimate Partner Violence and Substance Abuse in a Forensic Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Paul M.G.Emmelkamp, Prof. Dr. P.M.G. Emmelkamp, VU University of Amsterdam
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2008-KP-463
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Domestic Violence; Substance Abuse
Keywords: intimate partner violence; domestic violence; substance abuse; alcohol abuse; drug abuse; addiction
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- combined treatment (Experimental): A combined treatment containing cognitive behavioral therapy addressing partner violence and cognitive behavioral therapy addressing substance abuse
  Interventions: Behavioral: substance abuse/domestic violence treatment
- control condition (Active Comparator): Cognitive behavioral therapy addressing partner violence
  Interventions: Behavioral: CBT addressing partner violence

INTERVENTIONS:
Behavioral: substance abuse/domestic violence treatment — This intervention is comprised of 16 sessions of cognitive behavioral therapy. 8 sessions are addressing partner violence and 8 sessions are addressing substance abuse.
  Arms: combined treatment
Behavioral: CBT addressing partner violence — This treatment is comprised of 16 sessions of cognitive behavioral therapy addressing partner violence.
  Arms: control condition

SUMMARY:
Intimate partner violence is a significant societal problem. However, treatment of IPV perpetrators is far from effective, which may be partly due to the fact that the role of substance abuse is not taken into account. There is considerable evidence that a strong relationship between the use of alcohol and other drugs and intimate partner violence exists. Besides, a few studies indicate that reducing substance use may have a positive impact on IPV. Therefore, in this study, perpetrators of intimate partner violence with substance use disorders enrolled in domestic violence treatment will be randomly assigned to either standard treatment for offenders of domestic violence or a combination of the latter treatment with cognitive-behavioral therapy addressing substance abuse (combined treatment).

ELIGIBILITY:
Inclusion Criteria:

* A history of perpetration of intimate partner violence
* Current alcohol, cannabis and/or cocaine abuse or dependence
* Still in an intimate relationship with the victim

Exclusion Criteria:

* Not sufficient fluency in Dutch to complete treatment and measures
* (ab)use of crack cocaine and/or heroin
* In need of clinical detoxification
* Severe mental disorders, such as psychosis
* Severe cognitive disorders, such as Korsakoff's syndrome
* In treatment for other mental health problems
* Abuse of children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-09; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Quick Drinking Screen (QDS) | pretest, posttest, 6 & 12 months follow-up
Conflict Tactics Scale (CTS) | pretest, halfway treatment, posttest, 6 & 12 months follow-up
Timeline Followback interview | pretest, posttest
  Assesses daily substance use in the past 4 months

SECONDARY OUTCOMES:
Brief Symptom Inventory (BSI) | pretest, posttest, 6 and 12 moths follow-up
  Assesses general psychological complaints
Maudsly Marital Questionnaire (MMQ) | pretest, posttest, 6 and 12 months follow up
  Assesses marital satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Paul M.G. Emmelkamp, PhD., Principal Investigator — University of Amsterdam
Locations (1):
- De Waag Amsterdam & Rijnmond, Amsterdam / Rotterdam, Netherlands